CLINICAL TRIAL: NCT02141204
Title: Immunogenicity and Safety Study of Two Different Formulations of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine, Rotarix in Healthy Infants
Brief Title: Immunogenicity, Reactogenicity and Safety Study of Two Different Formulations of GSK Biologicals' Human Rotavirus Vaccine, Rotarix, in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116566; 2012-001875-35 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-10

CONDITIONS: Rotavirus
Keywords: Rotarix; HRV; Healthy infants; Liquid formulation; Lyophilized formulation; Human rotavirus vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV Liq Group (Experimental): Subjects aged 6 to 10 weeks at the time of first vaccination, who received two oral doses of Liquid Human Rotavirus Vaccine (HRV) according to a two-dose schedule, at Day 1 and Month 1.
  Interventions: Biological: HRV Liquid
- HRV Lyo Group (Active Comparator): Subjects aged 6 to 10 weeks at the time of first vaccination who received two oral doses of Lyophilized Human Rotavirus Vaccine (HRV) according to a two-dose schedule, at Day 1 and Month 1.
  Interventions: Biological: HRV Lyophilized

INTERVENTIONS:
Biological: HRV Liquid — Two doses administered orally according to a 0, 1-month schedule.
  Arms: HRV Liq Group
Biological: HRV Lyophilized — Two doses administered orally according to a 0, 1-month schedule.
  Arms: HRV Lyo Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, reactogenicity and safety of GSK Biologicals' HRV liquid vaccine compared to GSK Biologicals' HRV lyophilized vaccine when administered as a two-dose primary vaccination in healthy infants aged 6-10 weeks at dose one, with no previous history of rotavirus illness or vaccination.

While the lyophilized formulation of the HRV vaccine was licensed in India in February 2008, this study is conducted to generate additional clinical data for the liquid formulation of the HRV vaccine in India, as recommended by New Drug Advisory Committee on Vaccines (NDAC-Vaccines) of Drug Controller General of India (DCGI).

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/ Legally Acceptable Representative (s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/ LAR(s) of the subject prior to performing any study specific procedure.
* A male or female between, and including, 6 and 10 weeks of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Birth weight >2000 grams.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccine (Day-29 to Day 1), or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of any chronic drug therapy to be continued during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose of vaccine administration and ending at Visit 3; with the exception of the inactivated influenza vaccine, which is allowed at any time during the study, and other licensed routine childhood vaccinations, according to the local immunization practice.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of confirmed RV GE.
* Previous vaccination against RV.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, (including Severe Combined Immunodeficiency [SCID] disorder) based on medical history and physical examination.
* Uncorrected congenital malformation (such as Meckel's diverticulum) of the gastrointestinal tract that would predispose for Intussusception (IS).
* History of IS.
* Very prematurely born infants (born ≤28 weeks of gestation).
* Hypersensitivity to latex.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment. This warrants deferral of vaccination.

  * Fever is defined as temperature ≥38.0°C/100.4°F. The preferred location for measuring temperature in this study will be the oral cavity, the axilla or the rectum.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or medical history.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* GE within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 451 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- India (6):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vellore

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in India.
Pre-assignment Details: Out of 451 subjects enrolled in the study, 1 subject did not receive any study treatment and 1 vaccinated subject was eliminated from all analysis due to incorrect impartial witness.
  449 subjects were vaccinated and included in the Exposed Set, 419 subjects completed the study.
Period: Overall Study
Arm/Group | HRV Liq Group | HRV Lyo Group
Started | 224 | 225
Completed | 209 | 210
Not Completed | 15 | 15
Not completed — Lost to Follow-up | 2 | 1
Not completed — CONSENT WITHDRAWAL NOT DUE TO AE | 1 | 2
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 3 | 5
Not completed — NOT WILLING TO PARTICIPATE THIS VISIT | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRV Liq Group | HRV Lyo Group | Total
Number analyzed (Participants) | 224 | 225 | 449
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.8 (1.0) | 6.8 (1.1) | 6.8 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 120 | 220
  Male | 124 | 105 | 229
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 224 | 225 | 449

OUTCOME MEASURES:

1. Primary Outcome: Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibody Concentrations
Description: Serum anti-RV IgA antibody concentrations were expressed as geometric mean concentrations (GMCs).
Time Frame: At Month 2
Population: Analysis was performed on Per Protocol Set (PPS) for immunogenicity, which included all eligible subjects who received both doses of HRV vaccine, complied with vaccination schedule and for whom immunogenicity data were available at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | HRV Liq Group | HRV Lyo Group
Number analyzed (Participants) | 189 | 192
U/mL | 90.25 [67.28 to 121.06] | 94.16 [70.29 to 126.13]
Statistical Analysis 1: Comparison: HRV Liq Group vs HRV Lyo Group; Anti-RV IgA GMCs (non-inferiority): Non-inferiority comparison between GSK Biologicals' HRV liquid vaccine (HRV Liq Group) and GSK Biologicals' HRV lyophilized vaccine (HRV Lyo Group) in terms of geometric mean concentrations (GMCs) for anti-RV antibodies, one month after the administration of the second dose of study vaccine; Test type: Non-Inferiority — Lower limit (LL) of the two-sided 95% confidence interval (CI) for the ratio of anti-RV IgA antibody GMCs between HRV Liq Group over the HRV Lyo Group should be greater than or equal to (≥) 0.5; ANCOVA; 95% CI for the adjusted GMC ratio and the logarithm of baseline concentration were used as fixed effects in this ANCOVA model; GMC ratio = 0.93, 95% CI 2-sided [0.65 to 1.34]

2. Secondary Outcome: Percentage of Seroconverted Subjects for Anti-RV IgA Antibodies
Description: Seroconversion is defined as: - for subjects with a pre-vaccination anti-RV IgA antibody concentration lower than (<) 20 U/mL, seroconversion is achieved when the post-vaccination concentration is greater than or equal to (≥) 20 U/mL and
  - for subjects with a pre-vaccination anti-RV IgA antibody concentration ≥ 20 U/mL, seroconversion is achieved when the post-vaccination concentration is ≥ 2 times the pre-vaccination concentration.
Time Frame: At Month 2
Population: Analysis was performed on PPS for immunogenicity, which included all eligible subjects who received both doses of HRV vaccine, complied with vaccination schedule and for whom immunogenicity data were available at the specified time point.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HRV Liq Group | HRV Lyo Group
Number analyzed (Participants) | 189 | 192
Percentage of subjects | 54.5 [47.1 to 61.7] | 50.0 [42.7 to 57.3]

3. Secondary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs)
Description: Solicited general AEs assessed were fever (defined as temperature ≥ 38.0°C/100.4°F, the preferred location for measuring temperature in this study being the oral cavity, the axilla and the rectum), irritability/fussiness, diarrhea (defined as passage of three or more looser than normal stools within a day), vomiting (defined as one or more episodes of forceful emptying of partially digested stomach contents ≥1 hour after feeding within a day), loss of appetite and cough/runny nose. Any = occurrence of AE regardless of intensity grade or relation to study vaccination.
Time Frame: During the 8-day follow-up period after each vaccination (vaccines administered at Day 1 and Month 1)
Population: Analysis was performed on the Exposed Set (ES), which included all subjects with at least one study vaccine administration documented and with the diary card completed.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Liq Group | HRV Lyo Group
Number analyzed (Participants) | 224 | 225
Participants
  Cough/Runny Nose (Dose 1), Any | 22 | 24
  Cough/Runny Nose (Dose 2), Any: number analyzed (Participants) | 214 | 213
  Cough/Runny Nose (Dose 2), Any | 17 | 23
  Diarrhea (Dose 1), Any | 4 | 2
  Diarrhea (Dose 2), Any: number analyzed (Participants) | 214 | 213
  Diarrhea (Dose 2), Any | 3 | 3
  Fever (Dose 1), ≥ 38.0°C | 57 | 48
  Fever (Dose 2), ≥ 38.0°C: number analyzed (Participants) | 214 | 213
  Fever (Dose 2), ≥ 38.0°C | 50 | 53
  Irritability/Fussiness (Dose 1), Any | 71 | 83
  Irritability/Fussiness (Dose 2), Any: number analyzed (Participants) | 214 | 213
  Irritability/Fussiness (Dose 2), Any | 56 | 61
  Loss of appetite (Dose 1), Any | 33 | 42
  Loss of appetite (Dose 2), Any: number analyzed (Participants) | 214 | 213
  Loss of appetite (Dose 2), Any | 28 | 25
  Vomiting (Dose 1), Any | 22 | 22
  Vomiting (Dose 2), Any: number analyzed (Participants) | 214 | 213
  Vomiting (Dose 2), Any | 15 | 13

4. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE is defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, and reported in addition to those solicited during the clinical study and any 'solicited' AE with onset outside the specified period of follow-up for solicited AE. Any = occurrence of AE regardless of intensity grade or relation to study vaccination.
Time Frame: During the 31-day follow-up period across doses (vaccines administered at Day 1 and Month 1)
Population: Analysis was performed on the ES, which included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Liq Group | HRV Lyo Group
Number analyzed (Participants) | 224 | 225
Participants | 54 | 58

5. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed included any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization and/or resulted in disability/incapacity. Any = occurrence of SAE regardless of intensity grade or relation to study vaccination.
Time Frame: Throughout the study period (from Day 1 up to Month 2)
Population: Analysis was performed on the ES, which included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV Liq Group | HRV Lyo Group
Number analyzed (Participants) | 224 | 225
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 8-day (Day 1 to Day 8) follow-up period after each HRV vaccination. Unsolicited AEs: During the 31-day (Day 1 to Day 31) follow-up period after any HRV vaccination. SAEs: Throughout the study period (Day 1 to Month 2)
Arm/Group | HRV Liq Group | HRV Lyo Group
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/225
Serious Adverse Events (participants affected / at risk) | 7/224 | 2/225
Other Adverse Events (participants affected / at risk) | 146/224 | 162/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRV Liq Group (N=224) | HRV Lyo Group (N=225)
Bronchiolitis (Infections and infestations) | 3 (3) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRV Liq Group (N=224) | HRV Lyo Group (N=225)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 6 (8)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 33 (38) | 31 (38)
Crying (General disorders) | 1 (1) | 2 (2)
Injection site pain (General disorders) | 10 (12) | 7 (9)
Injection site swelling (General disorders) | 13 (17) | 12 (17)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 87 (119) | 91 (116)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (6)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 5 (5)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 44 (61) | 53 (68)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 87 (128) | 102 (144)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (44) | 47 (58)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT02141204/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT02141204/SAP_001.pdf